CLINICAL TRIAL: NCT06884098
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Bioequivalence of AD-228B with AD-2284 in Healthy Adult Volunteers
Brief Title: A Study to Compare PK Characteristics and Safety Profiles Between AD-228B and AD-2284
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-228BE-H
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Primary Hypercholesterolaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (RT) (Experimental): Period 1: Reference Drug (AD-2284), Period 2: Test Drug (AD-228B)
  Interventions: Drug: AD-228B; Drug: AD-2284
- Sequence B (TR) (Experimental): Period 1: Test Drug (AD-228B), Period 2: Reference Drug (AD-2284)
  Interventions: Drug: AD-228B; Drug: AD-2284

INTERVENTIONS:
Drug: AD-228B — AD-228B, 1Tab., Per Oral
Drug: AD-2284 — AD-2284, 1Tab., Per Oral

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-228B in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg (Female 45kg) and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Participation in other clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose (0hour) to 72hours
  Cmax of AD-228B
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose (0hour) to 72hours
  AUCt of AD-228B

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No